CLINICAL TRIAL: NCT06811753
Title: Impact of Robotic Surgery on Systemic Immune-inflammation Index in Gastric Cancer Patients
Brief Title: Impact of Robotic Surgery on Systemic Immune-inflammation Index
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: BasaksehirCamveSakura 2024-52
Record Dates: First submitted 2025-01-27; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; minimally invasive gastrectomy; systemic immune-inflammation index; Robotic surgery
MeSH Terms: conditions — Stomach Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: robotic surgery
  Interventions: Procedure: robotic surgery
- Group 2: laparoscopic surgery
- Group 3: open surgery

INTERVENTIONS:
Procedure: robotic surgery — minimally invasive surgery
  Groups: Group 1

SUMMARY:
Robotic surgery has been gaining attention because of the physical and metabolic morbidity of the conventional open technique.The systemic immune-inflammation index(SII) has emerged as a recent and more reliable biomarker.In our single-center retrospective cohort study, the investigators investigate SII in robotic gastrectomy in order to show the advantageous effect on immune system which the investigators think as the first study in the literature.

DETAILED DESCRIPTION:
Patients who underwent robotic gastrectomy between January 2021 and September 2024 were included in the study. The primary outcome was to ascertain the beneficial effects of robotic surgery in gastric cancer patients in terms of immune response. The secondary outcome was to examine the reliability of SII as a serum biomarker in comparison to previous studies on the diagnosis and postoperative follow-up of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

gastric cancer patients treated with surgery

Exclusion Criteria:

patients with haematologic malignancy, immune system disorder, antiplatelet drug usage, operations including splenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients operated for gastric cancer
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Systemic inflammatory index | One year
  Systemic inflammatory index (SII= (platelet count x neutrophil count)/lymphocyte count) was predicted to be lower in patients undergoing minimally invasive surgery. The neutrophil-lymphocyte ratio (NLR) and platelet lymphocyte ratio (PLT) have been the subject of investigation as potential biomarkers to show the immune response to the surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Yiğit Düzköylü, assoc. prof., Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Basakşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
demographics, surgery type, blood counts

REFERENCES:
- [Background] Lin GS, Huang XY, Lu J, Wu D, Zheng HL, Xu BB, Zheng CH, Li P, Xie JW, Wang JB, Lin JX, Chen QY, Cao LL, Lin M, Tu RH, Lin GT, Huang ZN, Lin JL, Huang CM. A good preoperative immune prognostic index is predictive of better long-term outcomes after laparoscopic gastrectomy compared with open gastrectomy for stage II gastric cancer in elderly patients. Surg Endosc. 2022 Mar;36(3):1814-1826. doi: 10.1007/s00464-021-08461-7. Epub 2021 Jun 2. PMID 34076769
- [Background] Zhu RH, Li PC, Zhang J, Song HH. Impact of minimally invasive surgery on immune function and stress response in gastric cancer patients. World J Gastrointest Surg. 2024 Aug 27;16(8):2484-2493. doi: 10.4240/wjgs.v16.i8.2484. PMID 39220065
- [Background] Aziz MH, Sideras K, Aziz NA, Mauff K, Haen R, Roos D, Saida L, Suker M, van der Harst E, Mieog JS, Bonsing BA, Klaver Y, Koerkamp BG, van Eijck CH. The Systemic-immune-inflammation Index Independently Predicts Survival and Recurrence in Resectable Pancreatic Cancer and its Prognostic Value Depends on Bilirubin Levels: A Retrospective Multicenter Cohort Study. Ann Surg. 2019 Jul;270(1):139-146. doi: 10.1097/SLA.0000000000002660. PMID 29334554
- [Background] Hirahara N, Matsubara T, Fujii Y, Kaji S, Kawabata Y, Hyakudomi R, Yamamoto T, Taniura T, Tajima Y. Comparison of the prognostic value of immunoinflammation-based biomarkers in patients with gastric cancer. Oncotarget. 2020 Jul 7;11(27):2625-2635. doi: 10.18632/oncotarget.27653. eCollection 2020 Jul 7. PMID 32676164
- [Background] Margraf A, Ludwig N, Zarbock A, Rossaint J. Systemic Inflammatory Response Syndrome After Surgery: Mechanisms and Protection. Anesth Analg. 2020 Dec;131(6):1693-1707. doi: 10.1213/ANE.0000000000005175. PMID 33186158
- [Background] Kinoshita T, Sato R, Akimoto E, Tanaka Y, Okayama T, Habu T. Reduction in postoperative complications by robotic surgery: a case-control study of robotic versus conventional laparoscopic surgery for gastric cancer. Surg Endosc. 2022 Mar;36(3):1989-1998. doi: 10.1007/s00464-021-08483-1. Epub 2021 Apr 12. PMID 33844086
- [Background] Nagata H, Kinoshita T, Komatsu M, Habu T, Yoshida M, Yura M. Comparison of robotic versus laparoscopic total gastrectomy for gastric cancer: A single-center retrospective cohort study in a Japanese high-volume center. Eur J Surg Oncol. 2024 Dec;50(12):108706. doi: 10.1016/j.ejso.2024.108706. Epub 2024 Sep 28. PMID 39357414